CLINICAL TRIAL: NCT06980519
Title: Treatment of Patients With Solid Tumor Cancers Via Intermediate-Size Patient Population Expanded Access Investigational New Drug (IND)
Brief Title: MNPR-101-PCTA-177Lu Expanded Access Program (EAP) for Patients With Solid Tumor Cancer
Status: Available | Type: Expanded Access
Sponsor: Monopar Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: IST-00Cb
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Solid Tumor; Solid Tumor Cancer; Oncology; uPAR-positive Solid Tumor; Urokinase Plasminogen Activator Receptor-positive Solid Tumor
Keywords: MNPR-101-PCTA-177Lu; SPECT; SPECT/CT; CT; Radiotherapy; Radiologic response; Single Photon Emission Computed Tomography; Computed Tomography; Monoclonal antibody radionuclide conjugate; Antibody radionuclide conjugate; Lutetium-177; Single Photon Emission Computed Tomography/Computed Tomography; Urokinase plasminogen activator receptor-positive; uPAR-positive; Positron emission tomography/computed tomography; PET/CT; EAP IST-00Ca
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: MNPR-101-PCTA-177Lu — MNPR-101-PCTA-177Lu is a monoclonal antibody-radionuclide conjugate intended to target and deliver radioactivity to solid tumors expressing uPAR.

SUMMARY:
The purpose of this Expanded Access Program (EAP) is to allow use of the investigational therapeutic agent, MNPR-101-PCTA-177Lu, for treatment of urokinase plasminogen activator receptor (uPAR)-positive solid tumors identified via positron emission tomography / computed tomography (PET/CT) with investigational imaging agent MNPR-101-DFO*-89Zr.

DETAILED DESCRIPTION:
This EAP will enroll patients with uPAR-positive solid tumor cancer confirmed by prior PET/CT imaging with MNPR-101-DFO*-89Zr (EAP IST-00Ca). Eligible patients will be treated with 1 cycle (as 2 fractionated doses) of investigational therapy, MNPR-101-PCTA-177Lu, at 1 of 4 planned dose levels. All enrolled patients will receive active treatment. Dosing of patients will begin at the lowest planned dose level. After 2 patients are dosed at a level, the next 2 patients may receive the next higher dose level, the same dose level, or a lower dose level, based upon the nature and severity of adverse reactions (side effects). The safety, tolerability, and potential antitumor effects (radiologic response) of MNPR-101-PCTA-177Lu will be evaluated over 12 weeks after dosing. The amount of radioactivity in blood samples will be checked over 4 weeks post dose. Patient survival will be followed up 6 months after the last dose received.

ELIGIBILITY:
Key Inclusion Criteria:

* Participated in the Expanded Access Program (EAP) IST-00Ca study
* Histologically or cytologically confirmed locally advanced or metastatic solid tumor cancer that is refractory to existing therapy(ies) known to provide clinical benefit, or for which no standard treatment is available, or is contraindicated
* Ability to understand and willingness to sign a written informed consent document

Key Exclusion Criteria:

* Chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy), or immunotherapy within 14 days prior to administration of MNPR-101-PCTA-177Lu
* Continuing ≥ Grade 3 adverse reactions from prior systemic therapy (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0)
* Prior treatment with any radiopharmaceutical or investigational agents within 4 weeks or 5 half-lives, whichever is longer, prior to administration of the first dose of MNPR-101-PCTA-177Lu other than MNPR-101-DFO*-89Zr
* Evidence of impaired organ function, particularly bone marrow, liver, kidney, or heart, according to specific test parameters
* Presence of other serious, non-malignant diseases or any other condition that, in the opinion of the investigator, could interfere with the objectives of the study, participant safety, or compliance

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim S. Delpassand, M.D. Chairman & Medical Director, Nuclear Medicine, Principal Investigator — Excel Diagnostics & Nuclear Oncology Center
Locations (1):
- Excel Diagnostics & Nuclear Oncology Center, Houston, Texas, United States